CLINICAL TRIAL: NCT00418964
Title: Functional, Clinical & Radiological Outcome of Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Control Clinical Trial Studies Comparing Bone Patella Bone, Single Bundle and Double Bundle Method.
Brief Title: Clinical Trial Comparing Three Anterior Cruciate Ligament Reconstructive Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Pauline Lui, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUHK00001
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Results first posted 2012-03-20 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Knee Injuries
Keywords: Anterior cruciate ligament rupture; Anterior cruciate ligament(A02.513.514.100)
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries | interventions — Bone-Patellar Tendon-Bone Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single bundle hamstring (Experimental)
  Interventions: Procedure: Single bundle hamstring
- Double bundle hamstring (Experimental)
  Interventions: Procedure: Double bundle hamstring
- Bone patellar tendon bone (Active Comparator)
  Interventions: Procedure: Bone patellar tendon bone

INTERVENTIONS:
Procedure: Single bundle hamstring — Single bundle hamstring
  Arms: Single bundle hamstring
Procedure: Double bundle hamstring — Double bundle hamstring
  Arms: Double bundle hamstring
Procedure: Bone patellar tendon bone — Bone patellar tendon bone
  Arms: Bone patellar tendon bone

SUMMARY:
The objective of this prospective study is to assess the clinical, functional and radiological outcomes of three different ACL reconstruction procedures: Bone Patella Bone graft, Single bundle hamstring graft and anatomical Double bundle graft in terms of pain, swelling, mobility, quadriceps girth size, stability, proprioception, bone mineral density and functional status.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) reconstruction surgery is one of the common procedures performed by orthopedic surgeons with approximately 100,000 cases performed per year in the United States. A large amount of sports injuries were related to ACL problem. As such, ACL injuries and treatment is still widely under intensive study.

Traditionally, ACL surgery has been focused on using bone patella bone graft and single bundle hamstring graft. Problems of knee pain, unstable fixation, rotational instability and degenerative changes were reported. Recently, the use of double bundle hamstring graft to reconstruct the ACL according its anatomy aiming to improve the rotational stability was proposed. However, results about the clinical, functional and radiological outcomes are limited.

The objective of this prospective pilot study is to assess the clinical, functional and radiological outcomes of three different ACL reconstruction procedures: Bone Patella Bone graft, Single bundle hamstring graft and anatomical Double bundle graft in terms of pain, swelling, mobility, quadriceps girth size, stability, proprioception, skin sensation, bone mineral density and functional status.

Subjects to be operated for ACL reconstruction and meeting the inclusion and exclusion criteria will be recruited. Subjects will be randomly assigned to the three surgical groups by block randomization. Demographic information, parameters in recovery domain, functional domain and stability domain, isokinetic test, motion analysis domain, proprioception and radiographical measurements will be made at baseline and at day 1, week 2, week 4, week 8, month 3, month 5, 1 year and 2 years post-surgery. The effect of different surgical techniques and time on the different outcomes will be analysed by 2-way ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Men above age 18-40 years old
* First ACL reconstruction surgery
* Single leg involvement

Exclusion Criteria:

* ACL injury less than 6 weeks as deleterious effect of the injury may affect the extension range
* Injury on Duty (IOD) cases
* Other associated injuries (Fractures, other ligaments involvement, neurovascular bundles injury),Chondral lesion with co-commitment intervention
* Concomitant meniscus repair in same operation, or within 3 months before the operation
* Significant OA changes
* Known chronic disease or receiving long term medications affecting bone metabolism, including anabolic steroids, medication for thyroid hormone therapy or osteoporosis
* Neurological deficit

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2006-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ming Chan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong SAR, China

RESULTS

PARTICIPANT FLOW:
Groups:
- HT-SB: Single bundle hamstring (hamstring autograft in a single bone tunnel)
- HT-DB: Double bundle hamstring (hamstring autograft in two bone tunnels)
- BPTB: Bone Patellar Tendon Bone (Bone patellar tendon bone autograft in a single bone tunnel)
Period: Overall Study
Arm/Group | HT-SB | HT-DB | BPTB
Started | 22 | 20 | 20
Completed | 21 | 17 | 14
Not Completed | 1 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HT-SB | HT-DB | BPTB | Total
Number analyzed (Participants) | 22 | 20 | 20 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 20 | 62
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.2 (5.0) | 26.4 (4.9) | 26.5 (5.0) | 25.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 22 | 20 | 20 | 62
Region of Enrollment [Number; unit: participants]
  China | 22 | 20 | 20 | 62

OUTCOME MEASURES:

1. Primary Outcome: International Knee Documentation Committee (IKDC)Knee Form 2000 Score
Description: It is a score on a scale from 0 to 100. It is a knee-specific measure of symptoms, function and sports activity of subjects based on self-report. 0 represents the worst while 100 represents the best score. The higher the score, the better the knee function.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HT-SB | HT-DB | BPTB
Number analyzed (Participants) | 21 | 17 | 14
Score on a scale | 85.7 (8.4) | 87.2 (12.8) | 84.6 (9.9)

2. Secondary Outcome: Percentage Distal Femoral Bone Mineral Density (BMD)Decrease
Description: % BMD decrease of distal femur of injured side with reference to the BMD at day 1 after surgery
Time Frame: 1 year
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: %

ADVERSE EVENTS:
Arm/Group | HT-SB | HT-DB | BPTB
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No